CLINICAL TRIAL: NCT00004070
Title: A Multi-Center, Open-Label, Multiple Administration, Rising Dose Study of the Safety, Tolerability, and Efficacy of IL-12 Gene Medicine in Patients With Unresectable or Recurrent/Refractory Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Gene Therapy in Treating Patients With Unresectable, Recurrent, or Refractory Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert I. Haddad, MD, Haddad, Robert MD, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99-081; P30CA006516 (NIH); VALENTIS-DFCI-99081; NCI-G99-1578; CDR0000067274 (Other: Other)
Record Dates: First submitted 1999-12-10; First posted 2004-06-04 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Head and Neck Cancer
Keywords: recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Interleukin-12; Interleukin-12 Subunit p35

STUDY DESIGN:
Intervention Model Description: This is a non-randomize phase I/II where patients are directly assigned treatment.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IL-12 Injection 3mg/ml [Phase I] (Experimental): The dosing schedule will consist of eight injections 3 mg/ml of formulated plasmid over a seven week period.
  Interventions: Biological: IL-12
- IL-12 Injection 6mg/ml [Phase I] (Experimental): The dosing schedule will consist of eight injections 6mg/ml of formulated plasmid over a seven week period.
  Interventions: Biological: IL-12
- IL-12 Injection MTD [Phase II] (Experimental): The dosing schedule will consist of eight injections over a seven week period of formulated plasmid at the MTD established in the phase I portion.
  Interventions: Biological: IL-12

INTERVENTIONS:
Biological: IL-12
  Other Names: NFSK; CLMF; P35; Interleukin-12 gene

SUMMARY:
Participant with squamous cell cancer of head and neck are invited to participate in this study. In this study the investigators will be Inserting the gene for interleukin-12 into a person's cancer cells with the anticipation to make the body build an immune response to kill more tumor cells.

DETAILED DESCRIPTION:
This is a Phase I/II trial to study the effectiveness of gene therapy in treating patients who have unresectable, recurrent, or refractory head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Females must be non-pregnant and non-lactating and either surgically sterile (via hysterectomy or bilateral tubal ligation), at least one year post-menopausal, or using acceptable methods of contraception for the duration of the study.
* Male subjects must be surgically sterile or using an acceptable method of contraception for the duration of the study.
* Disease: biopsy-proven unresectable or recurrent/refractory squamoussell_eareinoma_of_the:head-and-neck-(usualLy -Stage-Di-or-IV) -
* Tumor accessible to direct injection
* Karnofsky performance of at least 70%
* Life expectancy of at least three months
* Able to give written informed consent

Exclusion Criteria:

* Infection (concurrent or within previous 2 weeks)
* Active or clinically-relevant viral illnesses.
* Use of corticosteroids, high-dose non-steroidal antiinflammatory, or immunosuppressive drugs
* Chemotherapy, radiotherapy or immunotherapy within 28 days of study entry or during the course of study
* Respiratory disease sufficient to influence oxygenation of arterial blood
* Active liver disease with transaminases >3 times the upper limit of normal
* Previous history of liver disease
* NYHA Class EU or greater heart failure
* Serum creatinine of greater than 1.5 times the upper limit of normal
* Polymorphonuclear neutrophilic leukocyte count <3,000/mm3
* Platelet count <50,000/mm 3
* Tumor involving major blood vessels or obstructing the airway
* Previous treatment with viral-based gene therapy, recombinant DNA products, or bacterial plasmids
* Use of an investigational drug within 30 days of screening
* Other malignancies requiring treatment during the study
* Scheduled surgical resection
* History of autoimmune disease, including rheumatic disease, Crohn's disease, etc. ,
* Known allergy to polyvinylpyrrofidone (PVP) or related products
* History of psychiatric disabilities or seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 1999-07 (Actual); Primary Completion 2000-11 (Actual); Study Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) [Phase I] | Assessed during therapy up to 7 weeks.
  The MTD of IL-12 gene medicine is determined by the number of participants who experience a dose limiting toxicity (DLT). The MTD is defined as the highest dose at which fewer than one-third of patients experience a DLT. If no DLTs are observed in the two dose levels planned then evaluation of a third escalation will be considered. If the MTD is not reached, the dose selected for use in the phase II portion will be defined as the maximum volume that can be reasonably and safely injected into the tumor.
Dose Limiting Toxicity (DLT) [Phase I] | Assessed during therapy up to 7 weeks.
  A DLT was defined as grade 4 hematologic toxicity greater than 5 days duration or grade 3 or higher non-hematologic toxicity based on NCI common toxicity criteria (CTCAEv2).
Grade 3-4 Toxicity Rate [Phase II] | Assessed until last scheduled on-study visit up to visit 12/day 112.
  All Grade 3-4 events based on CTCAEv2 as reported on case report forms.

SECONDARY OUTCOMES:
Time to Progressive Disease (TTP) [Phase III] | Measurement by CT occurs up to the earliest of progression, death or 4 months after enrollment of last patient.
  Time to progression based on the Kaplan-Meier method is defined as the duration of time from study entry to documented first observation of progressive disease (PD).
  Time to progression based on the Kaplan-Meier method is defined as the duration of time from study entry to documented first observation of progressive disease (PD).
Response [Phase II] | Measurement by CT occurs up to visit 12/day 112.
  Best response on treatment classifies patients into 4 groups: complete response (CR) is complete disappearance of all signs, symptoms, biochemical and radiographic evidence of tumor for a minimum of 1 month; partial response (PR) is >/=50% decreases in tumor area for at least 4 weeks without an increase in size of other lesions of >25% or appearance of new lesions; progressive disease (PD) is >50% increase in size of any lesion present at baseline or after response, or appearance of a new lesion; and stable disease (SD) is neither PR or better nor PD.
Overall Survival (OS) [Phase II] | Measurement by CT occurs up to the earliest of progression, death or 4 months after enrollment of last patient.
  OS is defined as the duration of time from study entry to death or date last known alive and estimated using Kaplan-Meier (KM) methods.

CONTACTS AND LOCATIONS:
Overall Officials: A. Dimitrios Colevas, MD, Study Chair — NCI-Investigational Drug Branch
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No